CLINICAL TRIAL: NCT02625506
Title: Efficacy of Adding Tramadol as Adjunctive Analgesic With Levobupivacaine in Modified Pectoral Nerve Block for Modified Radical Mastectomy Surgery
Brief Title: Efficacy of Tramadol With Levobupivacaine for Modified Pectoral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R/15.05.67
Record Dates: First submitted 2015-11-21; First posted 2015-12-09 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Radical Mastectomy Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Levobupivacaine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine (Placebo Comparator): Patients will be subjected for radical mastectomy surgery and pectoral nerve block with levobupivacaine
  Interventions: Drug: Levobupivacaine
- Levobupivacaine and Tramadol (Active Comparator): Patients will be subjected for radical mastectomy surgery and pectoral nerve block with levobupivacaine and tramadol
  Interventions: Drug: Levobupivacaine and Tramadol

INTERVENTIONS:
Drug: Levobupivacaine — Ultrasound guided Pecs block will be performed using 20 ml of levobupivacaine
  Arms: Levobupivacaine
Drug: Levobupivacaine and Tramadol — Ultrasound guided Pecs block will be performed using 20 ml of levobupivacaine in conjunction with tramadol
  Arms: Levobupivacaine and Tramadol

SUMMARY:
The aim of this study is to evaluate the addition of tramadol combined with levobupivacaine in the reduction of postoperative pain, postoperative opioid consumption after modified radical mastectomy surgery.

DETAILED DESCRIPTION:
Breast surgeries are usually associated with sever postoperative pain ,good perioperative analgesic technique after breast surgery is always questionable Thoracic epidural and paravertebral blocks became the gold standard techniques for pain relief, however they may be associated with complications such as spinal cord injury, total spinal anesthesia ,inadvertent intravascular injection and pneumothorax.

Pecs block is less invasive procedure involving ultrasound guided inter-fascial injections which has been suggested as potential alternative analgesic technique.

The block produces excellent analgesia and can be used as a rescue block in cases where the analgesia provided by the paravertebral or epidural was patchy or ineffective .

Different drugs, including opioids, non-steroidal anti-inflammatory drugs, ketamine, clonidine, and neostigmine, have been added to local anesthetics to improve the duration and quality of analgesia.Tramadol has also been used for pain management of patients.

The power of this clinical trial was prospectively calculated using the G Power analysis program. Using a priory power analysis with accuracy mode calculations with visual analogue score (VAS) as the primary variant and assuming type I error protection of 0.05 and an effect size convention of 0.9, a total sample size of 54 patients (27 patients in each group) produced a power of 0.90. To protect against drop out cases we added 6 cases to the total number (total of 60 cases)

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II.
* Patients scheduled for radical mastectomy surgery.

Exclusion Criteria:

* Severe or uncompensated cardiovascular diseases
* renal diseases
* Hepatic diseases
* Endocrinal diseases.
* Pregnancy
* Postpartum
* Lactating females
* Allergy to study medications.
* Local skin infection
* Bleeding disorder
* Coagulation abnormality
* Spine deformity
* chest deformity
* Psychiatric disease

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | For the first 24 hours after surgery
  Postoperative pain will be assessed by utilizing visual analogue scale (VAS)

SECONDARY OUTCOMES:
Changes in heart rate | For one hour after surgery
Changes in blood pressure | For one hour after surgery
Changes in peripheral oxygen saturation | For one hour after surgery
Changes in end-tidal carbon dioxide tension | For one hour after surgery
Time for first analgesic request from extubation | for 24 hours after surgery
Total analgesics received for 24 hrs after surgery | for 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Salwa MS Hayes, MD, Principal Investigator — Assistant Professor of Anesthesia and Surgical Intensive Care; Reem A Sharkawy, MD, Study Director — Lecture of Anesthesia and Surgical Intensive Care; Tamer EM Farahat, MD, Study Chair — Lecture of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Mansoura Oncology Center, Al Mansurah, DK, Egypt